CLINICAL TRIAL: NCT04104867
Title: A Randomized Controlled Double-blinded of Effectiveness of Prokinetic Agents in Improving Abdominal Discomfort at Pre- and Post- Colonoscopy
Brief Title: Effectiveness of Prokinetic Agents in Improving Abdominal Discomfort at Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/524
Record Dates: First submitted 2019-09-17; First posted 2019-09-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — itopride; Domperidone

STUDY DESIGN:
Intervention Model Description: The participants will be randomly selected into one of the three arms (1:1:1 ratio) of a sealed, opaque envelope by one of the surgical residents or by the attending surgeon. The participants in each group will receive an envelope containing pills of identical appearance, each of Domperidone 10 mg, Itopride 50 mg or placebo. Both the attending physicians and the participants are blinded to the kind of study medication contained in the envelope.
  They are also informed to begin consuming the 3 liters of PEG-EL at 5.00 PM and complete it within 3 hours. Lastly, they are instructed to take the fourth pill at 6.00 AM on the day of colonoscopy. At the colonoscopy unit, the patients will be interviewed regarding the severity of abdominal discomfort during the preparation period after consuming the 3 liters of PEG-EL using a numeric pain rating scale.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Colonoscopy preparation by PEG-EL with Itopride (Active Comparator): Regular protocol for colonoscopy preparation, no solid foods are allowed except low residue diet during three days before the procedure. On the next day, only liquid diet consumption is allowed.On the day prior to colonoscopy, the patients can have only clear liquid and ad libitum throughout the day until midnight. They are also informed to begin consuming the 3 liters of PEG-EL at 5.00 PM and complete it within 3 hours one day befor colonoscopy.
  Interventions: Drug: Itopride
- Colonoscopy preparation by PEG-EL with Placebo (Placebo Comparator): Regular protocol for colonoscopy preparation, no solid foods are allowed except low residue diet during three days before the procedure. On the next day, only liquid diet consumption is allowed.On the day prior to colonoscopy, the patients can have only clear liquid and ad libitum throughout the day until midnight. They are also informed to begin consuming the 3 liters of PEG-EL at 5.00 PM and complete it within 3 hours one day befor colonoscopy.
  Interventions: Other: Placebo
- Colonoscopy preparation by PEG-EL with Domperidone (Active Comparator): Regular protocol for colonoscopy preparation, no solid foods are allowed except low residue diet during three days before the procedure. On the next day, only liquid diet consumption is allowed.On the day prior to colonoscopy, the patients can have only clear liquid and ad libitum throughout the day until midnight. They are also informed to begin consuming the 3 liters of PEG-EL at 5.00 PM and complete it within 3 hours one day befor colonoscopy.
  Interventions: Drug: Domperidone

INTERVENTIONS:
Drug: Itopride — the patients are instructed to take one pill of Itopride at 8.00 AM, 12.00 AM, 4.30 PM respectively before the dat of colonoscopy. Lastly, they are instructed to take the fourth pill at 6.00 AM on the day of colonoscopy.
  Other Names: Colonoscopy preparation by PEG-EL with Itopride
  Arms: Colonoscopy preparation by PEG-EL with Itopride
Drug: Domperidone — the patients are instructed to take one pill of Domperidone at 8.00 AM, 12.00 AM, 4.30 PM respectively before the dat of colonoscopy. Lastly, they are instructed to take the fourth pill at 6.00 AM on the day of colonoscopy.
  Other Names: Colonoscopy preparation by PEG-EL with Domperidone
  Arms: Colonoscopy preparation by PEG-EL with Domperidone
Other: Placebo — the patients are instructed to take one pill of placebo at 8.00 AM, 12.00 AM, 4.30 PM respectively before the dat of colonoscopy. Lastly, they are instructed to take the fourth pill at 6.00 AM on the day of colonoscopy.
  Other Names: Colonoscopy preparation by PEG-EL with Placebo
  Arms: Colonoscopy preparation by PEG-EL with Placebo

SUMMARY:
colonoscopy has been a preferred modality for colorectal screening which efficiently reduce in morbidity and mortality of the disaese. Although colonoscopy is a safe procedure, some patients may be suffered from major and minor complications. Abdominal discomfort (approximately 30%) usually persisted for 2 days after colonoscopy. These unsatisfactory experiences might affect the patients' willingness to return for a repeat colonoscopy, which the loss of adherence eventually reduce the effectiveness of colorectal cancer screening and surveillance.

Furthermore, during colonoscopy preparation, the patients are required to take large volume Polyethylene glycol-electrolyte lavage (PEG-EL) solution for bowel preparation which possibly lead to unpleasant gastrointestinal symptoms likewise.

Prokinetic agents are a class of drugs that promoted gastrointestinal motility and, thereby, decrease transit time. This stimulatory effect was considered clinically relevant to the management of disorders characterized by impaired motility, such as gastro-esophageal reflux, gastroparesis, intestinal pseudo-obstruction, and colonic inertia. Prokinetic agents have various mechanism such as Cholinergic agonists, Dopamine antagonists (i.e.Domperidone, Metoclopramide), Serotonergic agonists (i.e. Cisapride, Prucalopride,Mosapride). Interestingly, these drugs have been used to minimize the unpleasant abdominal symptoms from colonoscopy.

The objective of this study is to examine the efficacy of a prokinetic agent in alleviating abdominal discomfort during the period of colonoscopy preparation and aftercolonoscopy consecutively.

DETAILED DESCRIPTION:
The participants will be randomly selected into one of the three arms of this report's diagram (1:1:1 ratio) drawing of a sealed, opaque envelope by one of the surgical residents in charge or by the attending surgeon. The participants in each group will receive an envelope containing pills of identical appearance, each of Domperidone 10 mg, Itopride 50 mg or placebo. Both the attending physicians and the participants are blinded to the kind of study medication contained in the envelope.

From the regular protocol for colonoscopy preparation, no solid foods are allowed except low residue diet during three days before the procedure. On the next day, only liquid diet consumption is allowed. On the day prior to colonoscopy, the patients can have only clear liquid and ad libitum throughout the day until midnight. Additionally, the patients are instructed to take one pill at 8.00 AM, 12.00 AM, 4.30 PM respectively. They are also informed to begin consuming the 3 liters of PEG-EL at 5.00 PM and complete it within 3 hours. Lastly, they are instructed to take the fourth pill at 6.00 AM on the day of colonoscopy. At the colonoscopy unit, the patients will be interviewed regarding the severity of abdominal discomfort during the preparation period after consuming the 3 liters of PEG-EL using a 4-point scale (1=absent, 2=mild, 3=moderate, 4=severe). After finish the procedure, patients are informed to continue the study medication for three days consecutively.

The interviewer will make a phone call to the individuals at the first and third day after the procedure to confirm compliance of the study medication and inquiry about the severity of abdominal discomfort after procedure by using the same 4-point scale. If the patient can't be reached by a phone call or fail to continue the medication, this patient is classified as a drop out.

All data is collected by the main investigator from the patient chart and data recording form. Statistical analysis is performed using SPSS version 18. Patient characteristic and numerical data are reported by descriptive statistic such as mean, standard deviation. Parametric data is compared between groups using Chi-square, logistic regression analysis.Statistical significance is set at a level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are an outpatient scheduled for elective colonoscopy at Ramathibodi hospital
* Age between 18 to 80 years old
* American Society of Anesthesiologists (ASA) classification 1-2

Exclusion Criteria:

* Patients who reject to participate or withdrawal from the research
* History of Domperidone or Itopride allergy
* Patients who do not complete taking the study medication
* Patients who have ostomy or history of subtotal colectomy
* Patients who are diagnosed active colitis i.e. ulcerative colitis, TB colitis
* Take any pain reliever agent during the study period
* Patients who are unable to communicate comprehensibly
* Severe renal or hepatic impairment
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
abdominal pain | 24 hour
  the severity of abdominal pain using a 4-point scale (1=absent, 2=mild, 3=moderate, 4=severe)

SECONDARY OUTCOMES:
abdominal pain | 48 hour
  the severity of abdominal pain using a 4-point scale (1=absent, 2=mild, 3=moderate, 4=severe)
abdominal pain | 72 hour
  the severity of abdominal pain using a 4-point scale (1=absent, 2=mild, 3=moderate, 4=severe)

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quigley EMM. Prokinetics in the Management of Functional Gastrointestinal Disorders. Curr Gastroenterol Rep. 2017 Sep 8;19(10):53. doi: 10.1007/s11894-017-0593-6. PMID 28887755
- [Result] Panteris V, Haringsma J, Kuipers EJ. Colonoscopy perforation rate, mechanisms and outcome: from diagnostic to therapeutic colonoscopy. Endoscopy. 2009 Nov;41(11):941-51. doi: 10.1055/s-0029-1215179. Epub 2009 Oct 28. PMID 19866393
- [Result] de Jonge V, Sint Nicolaas J, van Baalen O, Brouwer JT, Stolk MF, Tang TJ, van Tilburg AJ, van Leerdam ME, Kuipers EJ; SCoPE consortium. The incidence of 30-day adverse events after colonoscopy among outpatients in the Netherlands. Am J Gastroenterol. 2012 Jun;107(6):878-84. doi: 10.1038/ajg.2012.40. Epub 2012 Mar 6. PMID 22391645
- [Result] Pignone M, Saha S, Hoerger T, Mandelblatt J. Cost-effectiveness analyses of colorectal cancer screening: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2002 Jul 16;137(2):96-104. doi: 10.7326/0003-4819-137-2-200207160-00007. PMID 12118964
- [Result] Mishima Y, Amano Y, Okita K, Takahashi Y, Moriyama N, Ishimura N, Furuta K, Ishihara S, Adachi K, Kinoshita Y. Efficacy of prokinetic agents in improving bowel preparation for colonoscopy. Digestion. 2008;77(3-4):166-72. doi: 10.1159/000141040. Epub 2008 Jun 25. PMID 18577886